CLINICAL TRIAL: NCT02923583
Title: A Randomized, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, and Immunogenicity of M834 (Abatacept Biosimilar Candidate), US-Sourced Orencia®, and European Union (EU)-Sourced Orencia® in Normal Healthy Volunteers
Brief Title: Assessment of Pharmacokinetics (PK) and Safety of M834 and Orencia ®, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Collaborators: Mylan Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MOM-M834-001
Record Dates: First submitted 2016-08-08; First posted 2016-10-04 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- M834 (Experimental): M834 (abatacept biosimilar candidate)
  Interventions: Biological: M834
- US Orencia® (Active Comparator): US-sourced Orencia® (abatacept)
  Interventions: Biological: US-Sourced Orencia®
- EU Orencia® (Active Comparator): EU-sourced Orencia® (abatacept)
  Interventions: Biological: EU-Sourced Orencia®

INTERVENTIONS:
Biological: M834
  Arms: M834
Biological: US-Sourced Orencia®
  Other Names: Abatacept
  Arms: US Orencia®
Biological: EU-Sourced Orencia®
  Other Names: Abatacept
  Arms: EU Orencia®

SUMMARY:
The purpose of this study is assess the pharmacokinetics and safety of M834 and Orencia ® following administration of a single-dose in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females 18 to 55 years of age, inclusive (of any ethnic origin).
2. Healthy as determined by medical history, physical examination, vital signs, and 12 lead electrocardiography (ECG) at screening.
3. Body mass index (BMI) between 18 and 32 kg/m2.
4. Body weight between 50.0 and 100.0 kg, inclusive.
5. Has smoked no more than 10 cigarettes, 3 cigars, or 3 pipes/day for at least 1 month prior to screening and is willing to comply with smoking restrictions during confinement at the study center.
6. Willing and able to comply with the requirements of the study.
7. Willing and able to sign a written informed consent.

Exclusion Criteria:

1. History and/or current presence of clinically significant angioedema, clinically significant hypersensitivity, or severe allergic reactions (either spontaneous or following drug administration), also including known or suspected clinically relevant drug hypersensitivity to any components of the study drugs or comparable drugs, or latex.
2. History of invasive systemic fungal infections (e.g., histoplasmosis, coccidioidomycosis) or other severe opportunistic infections; subjects with well-controlled or mild recurrent or chronic local fungal infections (e.g., tinea versicolor, onychomycosis, athlete's foot) may be included at the discretion of the Investigator.
3. A serious infection (associated with hospitalization and/or required intravenous anti-infectives) within 6 months of study drug administration or a significant infection requiring oral or topical anti-infectives within 4 weeks of study drug administration.
4. Any minor infection within 2 weeks of admission to the clinical unit on Day -1 that, in the opinion of the Investigator, may require systemic therapy or otherwise impact safety or participation in the study.
5. Herpes zoster infection in the last year or more than 1 herpes zoster infections in his/her lifetime.
6. Frequent chronic or recurrent infections (defined as >3 a year requiring prescribed antibiotic treatment; subjects with >3 viral upper respiratory infections may be considered based on Investigator discretion).
7. Previous administration of abatacept, belatacept, or biosimilar candidates referencing abatacept or belatacept.
8. Receipt of another recombinant human monoclonal antibody within 6 months prior to dosing in this trial, or within 5 half-lives, or within the expected period of pharmacodynamic effect; whichever is longest.
9. Intake of any study drug in another trial within 3 months prior to dosing in this trial or have received the last dose of an investigational drug >3 months ago but who are on extended follow-up, or planned dosing of an investigational drug (other than for this study) during the course of this trial.
10. History of alcohol abuse in the past year, or history of regular consumption of alcohol, or unwillingness to comply with the alcohol restrictions outlined.
11. History of drug abuse.
12. Donation of blood within 3 months or blood products (e.g., platelets within 6 weeks, plasma within 7 days) prior to dosing.
13. Use of any prescribed or non-prescribed medication, dietary supplements or herbal medication during the 2 weeks prior to dosing.
14. History of or current congestive heart failure.
15. History of or current signs or symptoms of demyelinating disease including optic neuritis and/or multiple sclerosis.
16. History of any cancer including lymphoma, leukemia, skin cancer and cervical carcinoma in situ.
17. History of immunodeficiency (including those subjects with a positive test for human immunodeficiency virus [HIV] I and II at screening) or other clinically significant immunological disorders, or auto-immune disorders. Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, metabolic, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders as judged by the investigator.
18. Received a live vaccine within 12 weeks prior to clinic admission (Day -1) or plan to receive a live vaccine during the study (up to and including Day 71).
19. Pregnant or breast-feeding women.
20. Men or women of childbearing potential who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include use of a condom with spermicide and one of the following highly effective methods: stable use of oral contraceptives or other prescription pharmaceutical contraceptive, intrauterine device (IUD); bilateral tubal ligation, vasectomy, additional barrier method [e.g., diaphragm, cap, sponge]).

    * Contraception is not required for subjects who are abstinent (abstinence should be their preferred and usual lifestyle; contraception should be used as described if subjects stop being abstinent), subjects in exclusive same-sex relationships, and post-menopausal females.

      * Postmenopausal women must be amenorrheic for at least 12 months, confirmed by follicle-stimulating hormone (FSH) level >40 IU/L at screening in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 243 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax) | Pre-dose; and post dose through day 85.
Area under the serum concentration (AUC) versus time curve from zero to last quantifiable concentration [AUC(0-last)] | Pre-dose; and post dose through day 85.
Area under the concentration-time curve in serum from time zero extrapolated to infinity [AUC(0-inf)] | Pre-dose; and post dose through day 85.

SECONDARY OUTCOMES:
The incidence of anti-drug antibodies (ADAs) | Pre-dose; and post dose through day 85.
Count and percentages of adverse events by treatment group. | Time of dosing up-to Day 85 post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Candida Fratazzi, MD, Study Director — Momenta Pharmaceuticals, Inc.; James Bush, MBChB, PhD, MRCS(Ed), MFPM, Principal Investigator — Covance Clinical Research Unit
Locations (2):
- United Kingdom (2):
  - Covance Clincal Research Unit Ltd, Leeds
  - Hammersmith Medicines Research (HMR), London

IPD SHARING:
Plan to Share IPD: Undecided